CLINICAL TRIAL: NCT07275905
Title: A Phase 1, Open-label, Randomized, Pilot and Feasibility Trial to Evaluate the Safety and Tolerability of the Achromobacter-targeting Bacteriophage Cocktail, AchromoPhage, Among Persons With Cystic Fibrosis and Chronic Achromobacter Lung Infections: The AchromoPhage Trial
Brief Title: Bacteriophages for Adults With Cystic Fibrosis and Chronic Achromobacter Lung Infection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ghady Haidar (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Ghady Haidar, Associate Professor of Medicine; Co-chair, Pittsburgh Phage Program (P3), University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25050049; 005199A123 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2025-11-24; First posted 2025-12-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis (CF); Achromobacter Infection
Keywords: Bacteriophage Therapy; Phage Therapy; AchromoPhage; Multidrug-Resistant Infections; Lung Infection; Pulmonary Infection; cystic fibrosis; Achromobacter
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Alone Arm (Experimental): Participants will receive a single weekly administration of AchromoPhage via the inhaled route for a total of three administrations. Each weekly administration consists of escalating inhaled doses of the cocktail:
  * Day 0 (visit 1, 1st week): 4×10⁷ total PFU
  * Day 7 (visit 2, 2nd week): 4×10⁸ total PFU
  * Day 14 (visit 3, 3rd week): 4×10⁹ total PFU
  Interventions: Biological: AchromoPhage
- Intravenous Alone Arm (Experimental): Participants will receive a single weekly administration of AchromoPhage via the intravenous route. Each weekly administration consists of escalating intravenous doses of the cocktail.
  * Day 0 (visit 1, 1st week): 4×10⁷ total PFU
  * Day 7 (visit 2, 2nd week): 4×10⁸ total PFU
  * Day 14 (visit 3, 3rd week): 4×10⁹ total PFU
  Interventions: Biological: AchromoPhage
- Combination Inhaled + Intravenous Arm (Experimental): Participants will receive a single weekly administration of AchromoPhage, which will consist of an inhaled dose followed by an intravenous dose given during the same study visit, with a 60-minute wait between doses. Weekly dose escalation will apply to each route, resulting in a total dose that is double that of the single route arms, as follows:
  * Day 0 (visit 1, 1st week): 8×10⁷ totalPFU [i.e. 4×10⁷ total PFU inhaled, followed by a 60-minute wait, then 4×10⁷ total PFU intravenous]
  * Day 7 (visit 2, 2nd week):8×10⁸ total PFU [i.e. 4×10⁸ total PFU inhaled, followed by a 60-minute wait, then 4×10⁸ total PFU intravenous]
  * Day 14 (visit 3, 3rd week): 8×10⁹ total PFU [i.e. 4×10⁹ total PFU inhaled, followed by a 60-minute wait, then 4×10⁹ total PFU intravenous]
  Interventions: Biological: AchromoPhage

INTERVENTIONS:
Biological: AchromoPhage — AchromoPhage is a cocktail of four genetically distinct, obligately lytic bacteriophages (phiACH01, phiACH04, phiACH06, phiACH07) with in vitro activity against >75% of a panel of 17 genetically diverse Achromobacter isolates from persons with cystic fibrosis. In this study, AchromoPhage will be administered by inhaled, intravenous, or sequential inhaled + intravenous routes with weekly dose escalation. Each participant will receive three weekly administrations, with escalating total doses of 4×10⁷ PFU, 4×10⁸ PFU, and 4×10⁹ PFU per route (double the total dose in the combination arm).
  Other Names: Phage; Bacteriophage

SUMMARY:
The goal of this clinical trial is to learn if a new treatment called AchromoPhage is safe and well tolerated in adults with cystic fibrosis (CF) who have long-term lung infections caused by Achromobacter bacteria. AchromoPhage is a mixture of four naturally occurring viruses, called phages, that are designed to target and kill Achromobacter.

This study will include 12 participants. People will be randomly assigned to one of three groups to receive AchromoPhage in different ways: by inhalation only, by intravenous (IV) infusion only, or by inhalation followed by IV infusion.

Participants will:

* Receive the study drug during clinic visits over a period of three weeks.
* Provide blood, sputum, nasal, and oral samples so researchers can measure how the phages move through the body, how long they stay, and whether the body develops a response against them.
* Complete breathing tests and quality-of-life questionnaires.

The main question this study will answer is whether AchromoPhage causes any serious or treatment-limiting side effects in the first 42 days after dosing. Researchers will also look at changes in lung function, quality of life, phage levels in the body, and how the treatment affects Achromobacter and other bacteria in the lungs.

The study is being run at the University of Pittsburgh (Pittsburgh, PA) and the University of California San Diego (San Diego, CA).

DETAILED DESCRIPTION:
AchromoPhage is a naturally derived bacteriophage cocktail composed of four genetically distinct, obligately lytic phages (phiACH01, phiACH04, phiACH06, and phiACH07) with demonstrated in vitro activity against Achromobacter species. The cocktail showed activity against more than 75% of a panel of 17 genetically diverse Achromobacter isolates collected from adults with cystic fibrosis. This study is designed to evaluate the safety and tolerability of AchromoPhage in adults with cystic fibrosis who have chronic Achromobacter lung infection.

This is an open-label, randomized Phase 1 pilot and feasibility trial conducted at two sites: the University of Pittsburgh, which will serve as the coordinating center, and the University of California San Diego. Eligible participants will be randomized to receive AchromoPhage by one of three delivery routes: inhaled administration, intravenous administration, or sequential inhaled followed by intravenous administration in the same visit. Each participant will receive three weekly administrations with escalating doses.

In addition to evaluating safety and tolerability, the trial will assess lung function and health-related quality of life, characterize pharmacokinetic profiles of AchromoPhage in blood and airway samples, and evaluate the humoral immune response to the administered phages. Exploratory analyses will examine pharmacodynamic effects, including changes in Achromobacter abundance, bacterial community profiles, antibiotic-phage interactions, and phage-pathogen dynamics.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Adults of any gender, age 18 years or greater at the time of enrollment.
  2. Weight of 40 kg or greater.
  3. Diagnosed with cystic fibrosis (CF).
  4. Stable respiratory symptoms within 30 days prior to screening.
  5. Chronic Achromobacter respiratory infection, defined as isolation by culture of Achromobacter species from two or more respiratory, oral, and/or nasopharyngeal samples provided by the participant within 24 months before the date of pre-screening.
  6. At least one Achromobacter isolate cultured from a respiratory, oral, and/or nasopharyngeal sample provided by the participant no more than 60 days before the date of planned enrollment must be susceptible to at least 1 phage in AchromoPhage cocktail using study assays.
  7. FEV1 ≥ (greater than or equal to) 40% of predicted at time of screening
  8. Ability and willingness to provide informed consent or, if applicable, the ability and willingness of legal guardian/representative to provide informed consent.
  9. Willingness to comply with study procedures.
  10. Ability to travel to the University of Pittsburgh or the University of California San Diego for phage administration and in-person visits.
  11. Agreement not to enroll in other bacteriophage studies or receive bacteriophages for clinical care during the study, except in life-saving situations.
  12. For females of reproductive potential, a negative urine pregnancy test at the time of consent (before randomization and dosing).
  13. Willingness to use highly effective contraception or other preventive measures to avoid conception during the study and for 6 months after the last phage dose.

Note, criteria 5 and 6 are the microbiologic criteria.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Serious medical illness requiring systemic treatment or hospitalization within 30 days prior to screening (unless medically stable and approved by the PI).
  2. Acute pulmonary exacerbation requiring systemic antibiotics within 30 days prior to screening.
  3. Acute respiratory illness, including viral infection, within 30 days prior to screening.
  4. Grade 3 or higher alanine aminotransferase (ALT) or aspartate aminotransferase (AST) at or within 30 days prior to screening, defined as ALT or AST values >5.0 x upper limit of normal (ULN).
  5. Currently breastfeeding, pregnant, or planning to become pregnant within 6 months.
  6. Hemoglobin < 8 g/dL
  7. Absolute neutrophil count < 1000 cells/uL
  8. Intolerance to inhaled therapies.
  9. Known allergy or sensitivity to components of the AchromoPhage cocktail.
  10. Any other condition that, in the PI's opinion, would interfere with the conduct of the study or would not be in the participant's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related Grade ≥4 adverse events or treatment-limiting toxicities | 42 Days
  Incidence of treatment-related Grade 4 or higher adverse events or any treatment-limiting toxicities, assessed overall and by treatment group, from the first dose through Day 42. Severity grading will follow the protocol-specified adverse event definitions.

SECONDARY OUTCOMES:
Change in health-related quality of life measured by the Cystic Fibrosis Questionnaire-(CFQ-R) | 42 Days
  Change in health-related quality of life from baseline to Day 42 measured using the Cystic Fibrosis Questionnaire-(CFQ-R), a validated, disease-specific instrument assessing physical, emotional, social, and respiratory health domains in cystic fibrosis.
  Construct measured: Health-related quality of life.
  Score range: Each domain generates a score from 0 to 100, where higher scores indicate better quality of life.
  Scoring: Domain scores are computed as linear transformations of raw responses; domains are not summed into a single composite score.
  Interpretation: Increases in domain scores represent improvement.
AchromoPhage Concentration by qPCR (Pharmacokinetic Outcome Measure) | Blood: Days 0, 7, 14, 21, 42. Sputum, nasal swabs, and oral swabs: Days 0, 7, 14, 21, 28, 35, and 42.
  Quantitative serum concentrations of each phage component of AchromoPhage will be measured by qPCR using primers that will amplify each of the 4 phages in the cocktail at predefined time points, following inhaled, intravenous, or combined administration.
  Blood PCR: Collected at 0-, 10-, 30-, 60-, 120-, 180-, and 240-minute intervals following AchromoPhage administration during dosing visits (Days 0, 7, and 14) and once on Days 21 and 42.
  Sputum, nasal swabs, and oral swabs: Collected weekly (Days 0, 7, 14, 21, 28, 35, and 42).
Number of Participants With Treatment-Emergent Serum Phage-Neutralizing Antibody Activity | Days 0, 7, 14, 21, 28, and 42
  Quantitative phage-neutralizing antibody activity will be measured in serum samples to assess treatment-emergent humoral immune responses following AchromoPhage administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ghady Haidar, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of California San Diego (UCSD), San Diego, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stellfox ME, Fernandes C, Shields RK, Haidar G, Hughes Kramer K, Dembinski E, Mangalea MR, Arya G, Canfield GS, Duerkop BA, Van Tyne D. Bacteriophage and antibiotic combination therapy for recurrent Enterococcus faecium bacteremia. mBio. 2024 Mar 13;15(3):e0339623. doi: 10.1128/mbio.03396-23. Epub 2024 Feb 14. PMID 38353560
- [Background] Haidar G, Chan BK, Cho ST, Hughes Kramer K, Nordstrom HR, Wallace NR, Stellfox ME, Holland M, Kline EG, Kozar JM, Kilaru SD, Pilewski JM, LiPuma JJ, Cooper VS, Shields RK, Van Tyne D. Phage therapy in a lung transplant recipient with cystic fibrosis infected with multidrug-resistant Burkholderia multivorans. Transpl Infect Dis. 2023 Apr;25(2):e14041. doi: 10.1111/tid.14041. Epub 2023 Mar 2. PMID 36864824
- [Background] Suh GA, Lodise TP, Tamma PD, Knisely JM, Alexander J, Aslam S, Barton KD, Bizzell E, Totten KMC, Campbell JL, Chan BK, Cunningham SA, Goodman KE, Greenwood-Quaintance KE, Harris AD, Hesse S, Maresso A, Nussenblatt V, Pride D, Rybak MJ, Sund Z, van Duin D, Van Tyne D, Patel R; Antibacterial Resistance Leadership Group. Considerations for the Use of Phage Therapy in Clinical Practice. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0207121. doi: 10.1128/AAC.02071-21. Epub 2022 Jan 18. PMID 35041506
- [Background] Schooley RT, Biswas B, Gill JJ, Hernandez-Morales A, Lancaster J, Lessor L, Barr JJ, Reed SL, Rohwer F, Benler S, Segall AM, Taplitz R, Smith DM, Kerr K, Kumaraswamy M, Nizet V, Lin L, McCauley MD, Strathdee SA, Benson CA, Pope RK, Leroux BM, Picel AC, Mateczun AJ, Cilwa KE, Regeimbal JM, Estrella LA, Wolfe DM, Henry MS, Quinones J, Salka S, Bishop-Lilly KA, Young R, Hamilton T. Development and Use of Personalized Bacteriophage-Based Therapeutic Cocktails To Treat a Patient with a Disseminated Resistant Acinetobacter baumannii Infection. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00954-17. doi: 10.1128/AAC.00954-17. Print 2017 Oct. PMID 28807909
- [Background] Tamma PD, Souli M, Billard M, Campbell J, Conrad D, Ellison DW, Evans B, Evans SR, Greenwood-Quaintance KE, Filippov AA, Geres HS, Hamasaki T, Komarow L, Nikolich MP, Lodise TP, Nayak SU, Norice-Tra C, Patel R, Pride D, Russell J, Van Tyne D, Chambers HF, FowlerJr VG, Schooley RT; Antibacterial Resistance Leadership Group. Safety and microbiological activity of phage therapy in persons with cystic fibrosis colonized with Pseudomonas aeruginosa: study protocol for a phase 1b/2, multicenter, randomized, double-blind, placebo-controlled trial. Trials. 2022 Dec 28;23(1):1057. doi: 10.1186/s13063-022-07047-5. PMID 36578069
- [Background] De Baets F, Schelstraete P, Van Daele S, Haerynck F, Vaneechoutte M. Achromobacter xylosoxidans in cystic fibrosis: prevalence and clinical relevance. J Cyst Fibros. 2007 Jan;6(1):75-8. doi: 10.1016/j.jcf.2006.05.011. Epub 2006 Jun 21. PMID 16793350
- [Background] Tetart M, Wallet F, Kyheng M, Leroy S, Perez T, Le Rouzic O, Wallaert B, Prevotat A. Impact of Achromobacter xylosoxidans isolation on the respiratory function of adult patients with cystic fibrosis. ERJ Open Res. 2019 Dec 8;5(4):00051-2019. doi: 10.1183/23120541.00051-2019. eCollection 2019 Oct. PMID 31832429
- [Background] Uyttebroek S, Chen B, Onsea J, Ruythooren F, Debaveye Y, Devolder D, Spriet I, Depypere M, Wagemans J, Lavigne R, Pirnay JP, Merabishvili M, De Munter P, Peetermans WE, Dupont L, Van Gerven L, Metsemakers WJ. Safety and efficacy of phage therapy in difficult-to-treat infections: a systematic review. Lancet Infect Dis. 2022 Aug;22(8):e208-e220. doi: 10.1016/S1473-3099(21)00612-5. Epub 2022 Mar 3. PMID 35248167